CLINICAL TRIAL: NCT07318935
Title: Examining the Impact of the Performing Arts on Hyperactivity, Impulsivity, and Inattention in Young Adults
Brief Title: Effects of Performing Arts on Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Julia Basso, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VT_IRB_23-811
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: ADHD
Keywords: electroencephalography; dance; exergaming; exercise; music; cognition; executive function; affective state; mood
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dance Exergaming (Experimental): Participants completed a 30-minute Just Dance exergaming session.
  Interventions: Behavioral: Dance Exergaming
- Stationary Cycling (Active Comparator): Participants completed a 30-minute stationary cycling session with matched audiovisual stimulation.
  Interventions: Behavioral: Stationary Cycling
- Music Listening (Active Comparator): Participants remained seated and listened to the matched song playlist while viewing Just Dance gameplay.
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Dance Exergaming — Participants in this intervention completed a dance-based exergaming session (Just Dance 2024) using the Nintendo Switch connected to a large projection screen. Each participant engaged in solo gameplay on Just Dance, following an on-screen coach through choreographed dance sequences set to selected songs. Only songs classified by the game developers as "Easy" were used to ensure consistent difficulty and exertion levels across participants. The total gameplay duration was 30 minutes. During the session, participants wore a Polar heart rate monitor to allow researchers to track physiological responses in real time.
  Arms: Dance Exergaming
Behavioral: Stationary Cycling — Participants in this intervention completed a stationary bike exercise session while listening to the same songs used in the dance exergaming condition. During biking, they watched prerecorded Just Dance gameplay videos to provide matched audiovisual stimulation across interventions. Before beginning the main session, participants performed a 3-minute self-paced warm-up and completed stretching as needed. Resistance on the bike was adjusted at the participant's preferred pace until they reached 50% of their age-predicted maximum heart rate, calculated as 220 minus age. Heart rate was continuously monitored using a Polar heart rate monitor to ensure they remained within the target training zone. Participants cycled for 30 minutes while listening to the randomized playlist.
  Arms: Stationary Cycling
Behavioral: Music Listening — Participants in this intervention remained seated and listened to the same songs used in the Just Dance intervention for approximately 30 minutes in a randomized order. During the session, they also watched prerecorded Just Dance gameplay videos to ensure visual stimulation matched across intervention conditions. During the session, participants wore a Polar heart rate monitor to allow researchers to track physiological responses in real time.
  Arms: Music Listening

SUMMARY:
This study examined whether dance-based video gaming could help young adults with Attention-Deficit/Hyperactivity Disorder (ADHD) improve attention, emotional wellbeing, and self-regulation. ADHD can affect focus, impulse control, coordination, and mood. Although medications are helpful for many individuals, they may produce side effects, may not lead to lasting improvement, or may not be accessible to everyone. Because of this, there has been growing interest in enjoyable, accessible, non-medication approaches to support symptom management. This research evaluated how different activities influenced the brain, body, and behavior. Participants were young adults ages 18-24 with a formal ADHD diagnosis. Each participant completed two visits: a baseline visit and an intervention visit. At baseline, participants completed questionnaires measuring ADHD symptoms, mood, and daily functioning. They also performed computer-based tasks assessing attention, inhibition, mental flexibility, and working memory while wearing an electroencephalography (EEG) cap to measure brain activity and a wearable heart rate monitor. Participants also completed balance assessments using a force plate that measured postural control. At the intervention visit, participants were randomly assigned to one of three 30-minute conditions:

* Dance exergaming (Just Dance video game) - active, dance-based movement
* Stationary biking - aerobic exercise while listening to music and watching dance gameplay videos
* Music listening - seated condition listening to the same music and watching the same videos

During these activities, EEG and heart rate were recorded. Afterward, participants repeated the same brain, cognitive, and balance assessments completed at baseline. A cool-down period was provided in all groups. This study allowed investigators to examine ADHD from multiple perspectives. The study assessed how movement, music, and dance influenced symptoms; how the brain responded during and after these activities; how the heart and nervous system adapted; and how balance and motor control changed. The study also evaluated how these systems (brain, body, and behavior) interacted with one another. By comparing dance exergaming with traditional aerobic exercise and a non-exercise condition, this study aimed to determine whether dance-based activity provided distinct benefits for young adults with ADHD. The goal was to better understand whether fun, creative, and widely accessible activities could support attention, emotional wellbeing, and physical regulation and whether they could complement existing treatment approaches.

DETAILED DESCRIPTION:
Participants were recruited from the greater Southwest Virginia and New River Valley regions through social media platforms (e.g., Facebook, Instagram, X), flyers distributed in the community, and in-person recruitment events. Interested individuals contacted the research team at embodiedbrainlab@gmail.com and were sent a brief screening questionnaire via REDCap along with an online screening consent form. Screening included the Physical Activity Readiness Questionnaire and questions assessing whether individuals had a formal ADHD diagnosis, relevant medical conditions or medications, and whether they met the study's age requirement (18-24 years). Individuals were also asked about exclusionary conditions such as neurological disorders, Tourette syndrome, epileptic disorders, and pregnancy. Those who met eligibility criteria were invited to review and sign the full informed consent form and were then asked to provide proof of their ADHD diagnosis, which was visually verified and retained in study files. Eligible participants were randomized to one of three intervention groups: a 30-minute dance exergaming session (experimental group), a 30-minute stationary biking session, or a 30-minute music-listening session (control groups). All study visits took place at the Science and Art of Movement Laboratory in the Center for the Arts at Virginia Tech.

Each participant completed two scheduled sessions. Availability was arranged through email or Microsoft Bookings, and participants were asked to abstain from caffeine on the day of testing due to its stimulant effects. The first visit served as a baseline assessment lasting approximately 90 minutes. During this session, participants completed questionnaires covering demographic information, medication use, recent food and drink intake, injury history, physical activity levels, and mental health constructs, including the Adult ADHD Self-Report Scale, Beck Depression Inventory, Beck Anxiety Inventory, and the DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure. Research staff then fitted participants with an EEG cap, after which participants completed a 5-minute resting-state recording of brain activity and heart rate while viewing a crosshair. Participants then performed four validated executive-function tasks on the INQUISIT platform-Color Word Stroop Task, Cued Go/No-Go Task, Wisconsin Card Sort Task, and Visual Digit Span Test-followed by six quiet-standing balance trials on a force plate (three with feet shoulder-width apart and three in tandem stance).

Approximately one week later, participants returned for their intervention session, which followed a parallel structure. They first completed the same questionnaire battery and resting EEG recording as during baseline. A 3-minute warm-up was completed prior to the assigned intervention. Participants then engaged in their randomized activity-dance exergaming, stationary biking, or music listening-for 30 minutes while wearing EEG and a Polar heart-rate monitor. Heart rate was continuously monitored, and research staff periodically checked in to ensure safety. Every 5 minutes, participants reported their perceived exertion using the Borg Rating of Perceived Exertion Scale. Following the intervention, all participants completed a 30-minute cool-down period with access to water, non-caffeinated tea, and comfortable seating. After cool-down, participants again completed a 5-minute resting EEG/heart rate recording, followed by the same executive-function and balance tasks they performed during the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 24
* Formal diagnosis of ADHD (inattentive, hyperactive-impulsive, or combined)

Exclusion Criteria:

* Current comorbid neurological disorder (e.g. seizure disorder; multiple sclerosis), tourette syndrome, or epileptic disorder
* Contraindication to physical activity
* Pregnancy
* Incarceration
* Inability to consent on own behalf
* Non-ambulatory

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
ADHD Symptom Severity | Within 1 week prior to and after invention
  Total score (0 to 72) on the Adult ADHD Self-Report Scale (ASRS) - v 1.1; higher scores indicate greater symptom severity

SECONDARY OUTCOMES:
Depression level | Within 1 week prior to and after invention
  Total score (0 to 63) on the Beck Depression Inventory II (BDI-II); higher scores indicate greater symptom severity
Anxiety level | Within 1 week prior to and after invention
  Total score (0-63) on the Beck Anxiety Inventory (BAI); higher scores indicate greater symptom severity
Attention | Within 1 week prior to and after invention
  Response time (ms) on the Stroop Color-Word Task for congruent and incongruent trials; lower values indicate faster/better response times
Inhibition | Within 1 week prior to and after invention
  Response time (ms) on the Go-/No-Go Task; lower values indicate faster/better response times
Inhibition | Within 1 week prior to and after intervention
  Percentage correct (%) on the Go-/No-Go Task; higher scores indicate better performance
Cognitive Flexibility | Within 1 week prior to and after invention
  Percentage correct (%) on Wisconsin Card Sorting Task; higher scores indicate better performance
Cognitive flexibility | Within 1 week prior to and after intervention
  Ability to learn task rules on Wisconsin Card Sorting Task (number or errors each time a new rule is introduced); positive score indicates improved performance whereas negative score indicates deteriorating performance
Working Memory | Within 1 week prior to and after invention
  Forward and backward recall (number of items recalled) on the Visual Digit Span Task; higher scores indicate better performance
Balance | Within 1 week prior to and after invention
  Force plate assessment in shoulder width and tandem stance measured via center of pressure (root mean square distance from the mean); higher values indicate lower stability
Balance | Within 1 week prior to and after intervention
  Force plate assessment in shoulder width and tandem stance measured via center of pressure (average velocity of the center of pressure); higher values indicate lower stability
Neural state during rest | Within 1 week prior to and after invention
  Power (log-transformed power in microvolts squared) in theta (4-8 hz), alpha (8-12 hz), beta (12-30 hz), and gamma (30-55 hz) frequency bands during a 5-minute resting baseline brain state; higher values indicate greater power
Neural state during cognitive tasks | Within 1 week prior to and after intervention
  Power (log-transformed power in microvolts squared) in theta (4-8 hz), alpha (8-12 hz), beta (12-30 hz), and gamma (30-55 hz) conducted during cognitive task assessment
Neural state during cognitive tasks | Within 1 week prior to and after intervention
  Amplitude of event-related potentials during cognitive tasks; higher value indicates a greater neural response to the task-stimulus - interpretation is component-specific
Neural state during cognitive tasks | Within 1 week prior to and after intervention
  Latency of event-related potentials during cognitive tasks; lower value indicates a faster neural response to the task-stimulus - interpretation is component-specific

OTHER OUTCOMES:
Sex | Within 1 week prior to intervention
  Sex at birth including female or male
Age | Within 1 week prior to intervention
  Age, ranging from 18 to 24
Race | Within 1 week prior to intervention
  Race including American Indian/Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, or more than one race/other
Ethnicity | Within 1 week prior to intervention
  Ethnicity including Hispanic/Latino or not Hispanic/Latino
Education level | Within 1 week prior to intervention
  Education level including finished high school or GED, some college, bachelor's degree, or advanced degree
Income level | Within 1 week prior to intervention
  Income level per year including under $15,000, $15,000 to $24,000, $25,000 to $34,999, $35,000 to $49,000, $50,000 to $74,999, $75,000 to $99,999, $100,000 to $149,000, $150,000 to $199,999, $200,000 or over, or don't know/not sure

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Basso, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified behavioral, physiological, and electroencephalography (EEG) data from this study will be shared. Data will be made available beginning 12 months after publication of the primary results and will remain accessible for 5 years. Qualified researchers may request access by submitting a brief proposal to the Principal Investigator outlining study aims and data security procedures. Approved researchers will sign a data use agreement. Only de-identified data will be provided, and use will be restricted to scientific, non-commercial purposes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available beginning 12 months after publication of the primary results and will remain accessible for 5 years.
Access Criteria: Qualified researchers may request access by submitting a brief proposal to the Principal Investigator outlining study aims and data security procedures. De-identified behavioral, physiological, and electroencephalography (EEG) data from this study will be shared.
URL: https://www.embodiedbrainlab.com/